CLINICAL TRIAL: NCT05828017
Title: Investigating Hearing Aid Frequency Response Curves 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sonova AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SRF-12972
Record Dates: First submitted 2023-03-24; First posted 2023-04-25 (Actual); Results first posted 2025-03-18 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2023-09

CONDITIONS: Hearing Loss, Sensorineural; Hearing Loss, Bilateral
Keywords: Hearing Loss; Hearing Aids; Frequency Response Curves
MeSH Terms: conditions — Hearing Loss, Sensorineural; Hearing Loss, Bilateral; Hearing Loss

STUDY DESIGN:
Intervention Model Description: The study is not a crossover study in it's true sense as there is only one arm. All participants will undergo all testing and will test each hearing aid variation. It should be noted that testing a different hearing aid variation (i.e., intervention) is done by simply clicking a button and having the hearing aid switch into a different variation. In this study, participants will go back and forth between different variations in order to make preference selections (Live Sound Quality or US Matrix Test task).
  Additionally, in other outcome measures, participants will listen to pre-recorded stimuli that have the various frequency response curves applied. In this case, participants once again will be exposed to different hearing aid curves while simply listening via headphones and making preference selections. In the end, participants can be exposed to different hearing aid variations (i.e., interventions) simultaneously and have the ability to go back and forth between interventions.
Masking Description: Participant were blinded to the type of intervention (i.e., hearing aid curve) or program they were comparing or rating. They were simply asked to specify which intervention they had a preference for.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Participants with Hearing Loss (Experimental): Individuals with hearing loss that meet the candidacy to wear hearing aids. All interventions are associated with the fitting of binaural hearing aids with various coupling methods. All participants will be assessed under all interventions.
  Interventions: Other: Hearing Aid - Standard Curve under Program 1; Device: Hearing Aid - Variation #1 under Program 1; Other: Hearing Aid - Variation #2 under Program 5 - Streaming Only; Other: Hearing Aid - Variation #3 under Program 5 - Streaming Only; Other: Hearing Aid - Variation #4under Program 5 - Streaming Only; Other: Hearing Aid - Standard Curve under Program 2; Other: Hearing Aid - Variation #1 under Program 2; Other: Hearing Aid - Standard Curve under Program 3; Other: Hearing Aid - Variation #1 under Program 3; Other: Hearing Aid - Standard Curve under Program 4; Other: Hearing Aid - Variation #1 under Program 4; Other: Unaided

INTERVENTIONS:
Other: Hearing Aid - Standard Curve under Program 1 — Our current hearing aids which will be programmed to our standard frequency response curve.
Device: Hearing Aid - Variation #1 under Program 1 — Hearing aids that will have the frequency response curve #1 adjusted and fit to the participant's hearing loss.
Other: Hearing Aid - Variation #2 under Program 5 - Streaming Only — Our current hearing aids which will be programmed to our standard frequency response curve.
Other: Hearing Aid - Variation #3 under Program 5 - Streaming Only — Hearing aids that will have the frequency response curve #3 adjusted and fit to the participant's hearing loss.
Other: Hearing Aid - Variation #4under Program 5 - Streaming Only — Hearing aids that will have the frequency response curve #4 adjusted and fit to the participant's hearing loss.
Other: Hearing Aid - Standard Curve under Program 2 — Our current hearing aids which will be programmed to our standard frequency response curve.
Other: Hearing Aid - Variation #1 under Program 2 — Hearing aids that will have the frequency response curve #1 adjusted and fit to the participant's hearing loss.
Other: Hearing Aid - Standard Curve under Program 3 — Our current hearing aids which will be programmed to our standard frequency response curve.
Other: Hearing Aid - Variation #1 under Program 3 — Hearing aids that will have the frequency response curve #1 adjusted and fit to the participant's hearing loss.
Other: Hearing Aid - Standard Curve under Program 4 — Our current hearing aids which will be programmed to our standard frequency response curve.
Other: Hearing Aid - Variation #1 under Program 4 — Hearing aids that will have the frequency response curve #1 adjusted and fit to the participant's hearing loss.
Other: Unaided — No hearing aids worn at all and participants tested as is.

SUMMARY:
Internal research on the manufacturer's hearing aid products has idenitfied areas in which the investigators can improve the hearing aid frequency response curve. Based on the conclusions of the first study, we have identified areas that require further analysis and testing prior to implementing of the proposed frequency response curve into our products. This study aims to investigate the current freqeuncy response curve in the manufacturer's products to variations of these curves to determine if hearing aid users prefer the variations over the manufacturer's standard curve.

DETAILED DESCRIPTION:
Internal testing has identified areas in which the investigators can improve the performance of the manufacturer's hearing aid products. This should potentially lead to increased hearing aid user satisfaction due to an improvement in sound quality and listener comfort. Therefore, a study is proposed in which hearing aid users will compare the manufacturer's current frequency response curve to variations made to the curve and determine which one they prefer while listening to live speech/music or while streaming speech/music and while in different listening enviroments.

ELIGIBILITY:
Inclusion Criteria:

* N3 - N5 Hearing losses
* Healthy Outer ear
* No visible congenital or traumatic deformity of the outer ear
* Symmetrical hearing loss - no air-bone gap greater than 10 dB at all 500, 1000, 2000, and 4000 Hz.
* Ability to answer questions and repeat sentences
* No history of problematic tinnitus or pain/discomfort from loud sounds
* No history of active drainage from the ears in the past 90 days
* Willingness to wear different styles of couplings
* Willingness to wear binaural fitting
* Experienced Users = more than 3 months of hearing aid experience
* Ability to travel to Sonova facilities

Exclusion Criteria:

* Contraindications to the medical device (MD) in this study (e.g. known hypersensitivity or allergy to the investigational products)
* Limited mobility/not able to come to the scheduled visit
* Inability to produce reliable hearing test results
* History of active drainage from the ear in the previous 90 days
* Abnormal appearance of the eardrum and ear canal.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-10-11 (Actual); Study Completion 2023-10-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jinyu Qian, PhD, Principal Investigator — Sonova AG
Locations (1):
- Sonova - Kitchener, Kitchener, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vaisberg J, Folkeard P, Levy S, Dundas D, Agrawal S, Scollie S. Sound Quality Ratings of Amplified Speech and Music Using a Direct Drive Hearing Aid: Effects of Bandwidth. Otol Neurotol. 2021 Feb 1;42(2):227-234. doi: 10.1097/MAO.0000000000002915. PMID 32976346
- [Background] Harianawala J, Galster J, Hornsby B. Psychometric Comparison of the Hearing in Noise Test and the American English Matrix Test. J Am Acad Audiol. 2019 Apr;30(4):315-326. doi: 10.3766/jaaa.17112. Epub 2018 Sep 25. PMID 30461418
- [Background] Wu YH, Stangl E, Chipara O, Hasan SS, Welhaven A, Oleson J. Characteristics of Real-World Signal to Noise Ratios and Speech Listening Situations of Older Adults With Mild to Moderate Hearing Loss. Ear Hear. 2018 Mar/Apr;39(2):293-304. doi: 10.1097/AUD.0000000000000486. PMID 29466265
- [Background] Neuman AC, Bakke MH, Hellman S, Levitt H. Effect of compression ratio in a slow-acting compression hearing aid: paired-comparison judgments of quality. J Acoust Soc Am. 1994 Sep;96(3):1471-8. doi: 10.1121/1.410289. PMID 7963011
- [Background] Caswell-Midwinter B, Whitmer WM. Discrimination of Gain Increments in Speech-Shaped Noises. Trends Hear. 2019 Jan-Dec;23:2331216518820220. doi: 10.1177/2331216518820220. PMID 30803400
- [Background] Smeds K, Wolters F, Rung M. Estimation of Signal-to-Noise Ratios in Realistic Sound Scenarios. J Am Acad Audiol. 2015 Feb;26(2):183-96. doi: 10.3766/jaaa.26.2.7. PMID 25690777
- [Background] Bisgaard N, Vlaming MS, Dahlquist M. Standard audiograms for the IEC 60118-15 measurement procedure. Trends Amplif. 2010 Jun;14(2):113-20. doi: 10.1177/1084713810379609. PMID 20724358

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was conducted via an internal database. Participants were recruited from May 2023 - October 2023. Participants were mainly contacted via email or telephone and only seen at the listed study locations.
Pre-assignment Details: All participants were exposed to all interventions. After enrollment and prior to testing, when applicable participant's hearing loss was assessed to confirm no significant changes from their baseline test. If a change in hearing loss was detected, it was evaluated to determine if the change was sufficient to place the participant outside the study's inclusion criteria. If so, the participant would be removed from the study.
Groups:
- Participants With Hearing Loss: Individuals with hearing loss that meet the candidacy to wear hearing aids. All interventions are associated with the fitting of binaural hearing aids with various coupling methods. All participants will be assessed under all interventions.
  Hearing Aid - Standard Curve: Our current hearing aids which will be programmed to our standard frequency response curve.
  Hearing Aid - Variation #1: Hearing aids that will have the frequency response curve adjusted and fit to the participant's hearing loss.
Period: Intake and Consent Form Completion
Arm/Group | Participants With Hearing Loss
Started | 25
Completed | 25
Not Completed | 0
Period: Review of Intake and Hearing Test Result
Arm/Group | Participants With Hearing Loss
Started | 25
Completed | 24
Not Completed | 1
Not completed — Removed by Investigator due to hearing loss change and no longer meeting study criteria. | 1
Period: Break Between Appointments 1 and 2
Arm/Group | Participants With Hearing Loss
Started | 24
Completed | 24
Not Completed | 0
Period: Live Sound Quality Ratings
Arm/Group | Participants With Hearing Loss
Started | 24
Completed | 24
Not Completed | 0
Period: Break Between Appointments 2 and 3
Arm/Group | Participants With Hearing Loss
Started | 24
Completed | 24
Not Completed | 0
Period: US Matrix Test Task
Arm/Group | Participants With Hearing Loss
Started | 24
Completed | 24
Not Completed | 0
Period: Streaming Sound Quality Ratings Task
Arm/Group | Participants With Hearing Loss
Started | 24
Completed | 24
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Participants With Hearing Loss
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 18
Age, Continuous [Mean (Full Range); unit: years] | 67.92 [26 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 11
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 25
Hearing Thresholds - PTA (500,1000,2000,4000 Hz) [Mean (Full Range); unit: Decibals in Hearing Level (dB HL)] — Hearing thresholds are measured via a hearing test. A hearing test is conducted by a licensed professional who is trained to conduct hearing tests and determine the severity of the hearing loss. Depending on the configuration and severity of the hearing loss dictates if a participant meets the requirements to join a clinical study. Hearing thresholds are measured across various frequencies and for both ears. The configuration of the hearing loss and average of 4 frequencies (500, 1000, 2000, and 4000 Hz (i.e., Pure Tone Average (PTA)) summarizes the severity of a participants hearing loss.
  Decibals in Hearing Level (dB HL) | 56 [39 to 92]

OUTCOME MEASURES:

1. Primary Outcome: Sound Quality Ratings - Listening Comfort - Program 1
Description: Participants will be asked to wear hearing aids and as they are exposed to listening environments. They will be asked to toggle between the two hearing aid programs (standard curve and variation #1) and determine which program provides increased listening comfort. Participants will be asked to make these ratings while seated in a sound booth.
  Scores will be tallied at the end to see which program of the two was preferred more in the different listening environments. Scores can range from 0 (the program was not preferred at all) to unlimited (dependent on the numbers of trials ran and samples tested). Higher scores will indicate that the program was preferred more than the other program and lowers scores mean the program was not preferred when compared to the other program.
Time Frame: 10 Minutes
Measure: Mean (Standard Deviation); unit: Mean Preference Counts per Participant
Arm/Group | Participants With Hearing Loss
Number analyzed (Participants) | 20
Mean Preference Counts per Participant
  Mean # of times Standard Curve was preferred in terms of listening comfort. | 4.78 (2.49)
  Mean # of times Variation #1 curve was preferred in terms of listening comfort. | 6.04 (2.16)
  Mean # of times there was no preference between the two curves in terms of listening comfort. | 2.36 (1.6)
Statistical Analysis 1: Comparison: Participants With Hearing Loss; This is to see if there is a difference in mean preference counts per participant between the standard curve, variation #1, and no preference counts; Test type: Superiority; p < 0.001, Chi-squared; Mean Difference (Final Values) = 1.107
Statistical Analysis 2: Comparison: Participants With Hearing Loss; This is to see if there is a difference between Variation #1 and the standard curve in terms of mean preference counts per participant; Test type: Superiority; p = 0.015, Chi-squared; Mean Difference (Final Values) = 0.544

2. Primary Outcome: Sound Quality Ratings - Overall Preference - Program 1
Description: Participants will be asked to wear hearing aids and as they are exposed to listening environments. They will be asked to toggle between the two hearing aid programs (standard curve and variation #1) and determine which program they prefer to listen to. Participants will be asked to make these ratings while seated in a sound booth.
  Scores will be tallied at the end to see which program of the two was preferred more in the different listening environments. Scores can range from 0 (the program was not preferred at all) to unlimited (dependent on the numbers of trials run and samples tested). Higher scores will indicate that the program was preferred more than the other program and lowers scores mean the program was not preferred when compared to the other program.
Time Frame: 10 Minutes
Measure: Mean (Standard Deviation); unit: Mean Preference Counts per Participant
Arm/Group | Participants With Hearing Loss
Number analyzed (Participants) | 20
Mean Preference Counts per Participant
  Mean # of times Standard Curve was preferred in terms of overall preference. | 4.83 (2.62)
  Mean # of times Variation #1 curve was preferred in terms of overall preference. | 5.85 (2.28)
  Mean # of times there was no preference between the two curves in terms of overall preference. | 2.33 (1.76)
Statistical Analysis 1: Comparison: Participants With Hearing Loss; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.001, Chi-squared; Mean Difference (Final Values) = 1.039
Statistical Analysis 2: Comparison: Participants With Hearing Loss; This is to see if there is a difference in mean preference counts between the standard curve and variation #1; Test type: Superiority; p = 0.03569, Chi-squared; Mean Difference (Final Values) = 0.47

3. Primary Outcome: Sound Quality Ratings - Speech Clarity - Program 1
Description: Participants will be asked to wear hearing aids and as they are exposed to listening environments. They will be asked to toggle between the two hearing aid programs (standard curve and variation #1) and determine which program has better speech clarity. Participants will be asked to make these ratings while seated in a sound booth.
  Scores will be tallied at the end to see which program of the two was preferred more in the different listening environments. Scores can range from 0 (the program was not preferred at all) to unlimited (dependent on the numbers of trials ran and samples tested). Higher scores will indicate that the program was preferred more than the other program and lowers scores mean the program was not preferred when compared to the other program.
Time Frame: 10 minutes
Measure: Mean (Standard Deviation); unit: Mean Preference Counts per Participant
Arm/Group | Participants With Hearing Loss
Number analyzed (Participants) | 20
Mean Preference Counts per Participant
  Mean # of times Standard Curve was preferred in terms of speech clarity | 3.24 (1.56)
  Mean # of times Variation #1 was preferred in terms of speech clarity | 3.00 (1.27)
  Mean # of times there was no preference between the two curves in terms of speech clarity | 2.73 (1.8)
Statistical Analysis 1: Comparison: Participants With Hearing Loss; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.069, Chi-squared; Mean Difference (Final Values) = 0.365
Statistical Analysis 2: Comparison: Participants With Hearing Loss; This is to see if there is a difference in mean preference counts between the standard curve and variation #1; Test type: Superiority; p = 0.6976, Chi-squared; Mean Difference (Final Values) = 0.087

4. Primary Outcome: Sound Quality Ratings - Noise Intrusion - Program 1
Description: Participants will be asked to wear hearing aids and as they are exposed to listening environments. They will be asked to toggle between the two hearing aid programs (Standard curve and variation #1) and determine which program has more noise intrusion. Participants will be asked to make these ratings while seated in a sound booth.
  Scores will be tallied at the end to see which program of the two was preferred more in the different listening environments. Scores can range from 0 (the program was not preferred at all) to unlimited (dependent on the numbers of trials ran and samples tested). Higher scores will indicate that the program was preferred more than the other program and lowers scores mean the program was not preferred when compared to the other program.
Time Frame: 10 Minutes
Measure: Mean (Standard Deviation); unit: Mean Preference Counts per Participant
Arm/Group | Participants With Hearing Loss
Number analyzed (Participants) | 20
Mean Preference Counts per Participant
  Mean # of times Standard Curve was preferred in terms of noise intrusion | 3.84 (2.81)
  Mean # of times variation #1 was preferred in terms of noise intrusion | 6.21 (2.18)
  Mean # of times there was no preference between the two curves in terms of noise intrusion | 2.72 (1.41)
Statistical Analysis 1: Comparison: Participants With Hearing Loss; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.001, Chi-squared; Mean Difference (Final Values) = 0.876
Statistical Analysis 2: Comparison: Participants With Hearing Loss; This is to see if there is a difference in mean preference counts between the standard curve and variation #1; Test type: Superiority; p = 0.0013, Chi-squared; Mean Difference (Final Values) = 0.728

5. Primary Outcome: Sound Quality Ratings - Listening Comfort - Program 2
Description: as for outcome 1
Time Frame: 10 Minutes
Measure: Mean (Standard Deviation); unit: Mean Preference Counts per Participant
Arm/Group | Participants With Hearing Loss
Number analyzed (Participants) | 20
Mean Preference Counts per Participant
  Mean # of times Standard Curve was preferred in terms of listening comfort. | 1.55 (0.82)
  Mean # of times Variation #1 curve was preferred in terms of listening comfort. | 1.71 (0.726)
  Mean # of times there was no preference between the two curves in terms of listening comfort. | 1.46 (0.519)
Statistical Analysis 1: Comparison: Participants With Hearing Loss; This is to see if there is a difference in mean counts per participant between the standard curve, variation #1, and no preference counts; Test type: Superiority; p = 0.522, Chi-squared; Mean Difference (Final Values) = 0.18
Statistical Analysis 2: Comparison: Participants With Hearing Loss; This is to see if there is a difference in mean counts between the standard curve and variation #1; Test type: Superiority; p = 0.27, Chi-squared; Mean Difference (Final Values) = 0.24

6. Primary Outcome: Sound Quality Ratings - Overall Preference - Program 2
Description: as for outcome 2
Time Frame: 10 Minutes
Measure: Mean (Standard Deviation); unit: Mean Preference Counts per Participant
Arm/Group | Participants With Hearing Loss
Number analyzed (Participants) | 20
Mean Preference Counts per Participant
  Mean # of times Standard Curve was preferred in terms of overall preference. | 1.5 (0.85)
  Mean # of times Variation #1 curve was preferred in terms of overall preference. | 1.79 (0.69)
  Mean # of times there was no preference between the two curves in terms of overall preference. | 1.54 (0.66)
Statistical Analysis 1: Comparison: Participants With Hearing Loss; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.28, Chi-squared; Mean Difference (Final Values) = 0.25
Statistical Analysis 2: Comparison: Participants With Hearing Loss; This is to see if there is a difference in mean counts per participant between the standard curve and variation #1; Test type: Superiority; p = 0.11, Chi-squared; Mean Difference (Final Values) = 0.35

7. Primary Outcome: Sound Quality Ratings - Noise Intrusion - Program 2
Description: as for outcome 4
Time Frame: 10 Minutes
Measure: Mean (Standard Deviation); unit: Mean Preference Counts per Participant
Arm/Group | Participants With Hearing Loss
Number analyzed (Participants) | 20
Mean Preference Counts per Participant
  Mean # of times Standard Curve was preferred in terms of noise intrusion | 1.45 (0.82)
  Mean # of times variation #1 was preferred in terms of noise intrusion | 1.77 (0.83)
  Mean # of times there was no preference between the two curves in terms of noise intrusion | 1.5 (0.52)
Statistical Analysis 1: Comparison: Participants With Hearing Loss; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.52, Chi-squared; Mean Difference (Final Values) = 0.18
Statistical Analysis 2: Comparison: Participants With Hearing Loss; This is to see if there is a difference in mean counts per participant between the standard curve and variation #1; Test type: Superiority; p = 0.26, Chi-squared; Mean Difference (Final Values) = 0.25

8. Primary Outcome: Sound Quality Ratings - Listening Comfort - Program 3
Description: as for outcome 1
Time Frame: 10 Minutes
Measure: Mean (Standard Deviation); unit: Mean Preference Counts per Participant
Arm/Group | Participants With Hearing Loss
Number analyzed (Participants) | 20
Mean Preference Counts per Participant
  Mean # of times Standard Curve was preferred in terms of listening comfort. | 1.73 (0.79)
  Mean # of times Variation #1 curve was preferred in terms of listening comfort. | 1.54 (0.66)
  Mean # of times there was no preference between the two curves in terms of listening comfort. | 2.00 (1.00)
Statistical Analysis 1: Comparison: Participants With Hearing Loss; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.16, Chi-squared; Mean Difference (Final Values) = 0.3
Statistical Analysis 2: Comparison: Participants With Hearing Loss; This is to see if there is a difference in mean counts per participant between the standard curve and variation #1; Test type: Superiority; p = 0.37, Chi-squared; Mean Difference (Final Values) = 0.19

9. Primary Outcome: Sound Quality Ratings - Overall Preference - Program 3
Description: as for outcome 2
Time Frame: 10 Minutes
Measure: Mean (Standard Deviation); unit: Mean Preference Counts per Participant
Arm/Group | Participants With Hearing Loss
Number analyzed (Participants) | 20
Mean Preference Counts per Participant
  Mean # of times Standard Curve was preferred in terms of overall preference. | 1.80 (0.77)
  Mean # of times Variation #1 curve was preferred in terms of overall preference. | 1.54 (0.66)
  Mean # of times there was no preference between the two curves in terms of overall preference. | 2.17 (0.98)
Statistical Analysis 1: Comparison: Participants With Hearing Loss; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.08, Chi-squared; Mean Difference (Final Values) = 0.35
Statistical Analysis 2: Comparison: Participants With Hearing Loss; This is to see if there is a difference in mean counts per participant between the standard curve and variation #1; Test type: Superiority; p = 0.31, Chi-squared; Mean Difference (Final Values) = 0.22

10. Primary Outcome: Sound Quality Ratings - Speech Clarity - Program 3
Description: as for outcome 3
Time Frame: 10 minutes
Measure: Mean (Standard Deviation); unit: Mean Preference Counts per Participant
Arm/Group | Participants With Hearing Loss
Number analyzed (Participants) | 20
Mean Preference Counts per Participant
  Mean # of times Standard Curve was preferred in terms of speech clarity | 1.73 (0.79)
  Mean # of times Variation #1 was preferred in terms of speech clarity | 1.67 (0.70)
  Mean # of times there was no preference between the two curves in terms of speech clarity | 1.90 (0.87)
Statistical Analysis 1: Comparison: Participants With Hearing Loss; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.21, Chi-squared; Mean Difference (Final Values) = 0.27
Statistical Analysis 2: Comparison: Participants With Hearing Loss; This is to see if there is a difference in mean counts per participant between the standard curve and variation #1; Test type: Superiority; p = 0.085, Chi-squared; Mean Difference (Final Values) = 0.38

11. Primary Outcome: Sound Quality Ratings - Noise Intrusion - Program 3
Description: as for outcome 4
Time Frame: 10 Minutes
Measure: Mean (Standard Deviation); unit: Mean Preference Counts per Participant
Arm/Group | Participants With Hearing Loss
Number analyzed (Participants) | 20
Mean Preference Counts per Participant
  Mean # of times Standard Curve was preferred in terms of noise intrusion | 1.75 (0.75)
  Mean # of times variation #1 was preferred in terms of noise intrusion | 1.50 (0.65)
  Mean # of times there was no preference between the two curves in terms of noise intrusion | 1.64 (0.81)
Statistical Analysis 1: Comparison: Participants With Hearing Loss; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.86, Chi-squared; Mean Difference (Final Values) = 0.08
Statistical Analysis 2: Comparison: Participants With Hearing Loss; This is to see if there is a difference in mean counts per participant between the standard curve and variation #1; Test type: Superiority; p = 1, Chi-squared; Mean Difference (Final Values) = 0

12. Primary Outcome: Sound Quality Ratings - Overall Preference - Program 4
Description: as for outcome 2
Time Frame: 10 Minutes
Measure: Mean (Standard Deviation); unit: Mean Preference Counts per Participant
Arm/Group | Participants With Hearing Loss
Number analyzed (Participants) | 20
Mean Preference Counts per Participant
  Mean # of times Standard Curve was preferred in terms of overall preference. | 1.30 (0.83)
  Mean # of times Variation #1 curve was preferred in terms of overall preference. | 1.60 (0.51)
  Mean # of times there was no preference between the two curves in terms of overall preference. | 1.94 (0.92)
Statistical Analysis 1: Comparison: Participants With Hearing Loss; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.009, Chi-squared; Mean Difference (Final Values) = 0.607
Statistical Analysis 2: Comparison: Participants With Hearing Loss; This is to see if there is a difference in mean counts per participant between the standard curve and variation #1; Test type: Superiority; p = 0.61, Chi-squared; Mean Difference (Final Values) = 0.30

13. Secondary Outcome: US Matrix Test in Noise Results - dB SNR 50%
Description: Oldenburg Sentence Test (OLSA) sentences were presented to participants while they were aided under the standard curve, aided under variation #1 frequency response curve, and unaided.
  Participants are presented with sentences from a loudspeaker placed Infront of them and noise from 7 loudspeakers placed around them (8 speakers placed 30 degrees apart from each other). Participants were asked to repeat what they heard. Correct repetition results in the next sentence to be presented at a lower sound level. Incorrect repetition results in an increase in presentation level for the next sentence. 20 sentences are presented for each condition (i.e., unaided, aided with the standard curve, and aided with the proposed frequency response curve). decibel signal to noise ratio (dB SNR) at 50% correctness scores were calculated at the end and compared amongst the three conditions. There are no minimum or maximum values, however lower scores indicate better performance.
Time Frame: 30 Minutes
Population: 1 participants data was removed as they were not accurate in their response and the US Matrix test software could not accurately measure their SRT50 score although mutliple attempts were made.
Measure: Mean (Standard Deviation); unit: dB SNR - (units on a scale)
Arm/Group | Participants With Hearing Loss
Number analyzed (Participants) | 19
dB SNR - (units on a scale)
  Hearing Aid - Variation # 1 - Mean SRT50% Score | -4.69 (2.35)
  Hearing Aid - Standard Curve - Mean SRT50% Score | -5.38 (2.15)
  Hearing Aid - Unaided - Mean SRT50% Score | -0.85 (4.7)
Statistical Analysis 1: Comparison: Participants With Hearing Loss; This is to see if there is a difference in mean SRT50 scores between the standard curve, variation #1, and no preference counts; Test type: Superiority; p < 0.001, ANOVA; Mean Difference (Final Values) = 0.28, 95% CI 2-sided [0.11 to 1.00]
Statistical Analysis 2: Comparison: Participants With Hearing Loss; This is to see if there is a difference in SRT 50 scores between the standard curve and variation #1; Test type: Superiority; p = 0.357, ANOVA; Mean Difference (Final Values) = 0.02, 95% CI 2-sided [0 to 1]

14. Secondary Outcome: Sound Quality Ratings - Streaming
Description: Participants will be asked to listen to various streamed stimuli via headphones. They will be asked to toggle between three programs (standard curve, variation #2, and variation #3) and determine which one they prefer the most, which one the prefer the least, and which one they prefer in the middle. Participants will be asked to make these ratings while seated in a sound booth.
  Scores will be tallied at the end to see which program was constantly the most preferred across the various stimuli. Highers rankings will indicate that the program was preferred more than the other program and lower rankings mean the program was not preferred when compared to the other program.
Time Frame: 1 hour
Measure: Number; unit: Ratings
Arm/Group | Participants With Hearing Loss
Number analyzed (Participants) | 20
Ratings
  Count of times Variation # 2 was rated the highest. | 120
  Count of times Variation #3 was rated the highest. | 119
  Count of times Variation #4 was rated the highest | 65
  Count of times Variation #2 was rated in the middle. | 56
  Count of times Variation #3 was rated in the middle. | 83
  Count of times Variation #4 was rated in the middle. | 89
  Count of times Variation #2 was rated the lowest. | 128
  Count of times Variation #3 was rated the lowest. | 102
  Count of times Variation #4 was rated the lowest. | 74
Statistical Analysis 1: Comparison: Participants With Hearing Loss; This is to see if there is a difference in most preferred program counts between variations #2, #3, and #4; Test type: Superiority; p < 0.01, Chi-squared; Total Count - Cramer's V = 0.7
Statistical Analysis 2: Comparison: Participants With Hearing Loss; This is to see if there is a difference in most preferred program counts between variations #2 and #3; Test type: Superiority; p = 0.94, Chi-squared; Total Count - Cramer's V = 0.01
Statistical Analysis 3: Comparison: Participants With Hearing Loss; This is to see if there is a difference in most preferred program counts between variations #2 and #4; Test type: Superiority; p = 0.94, Chi-squared; Total Count - Cramer's V = 0.014
Statistical Analysis 4: Comparison: Participants With Hearing Loss; This is to see if there is a difference in somewhat preferred (i.e. rated in the middle) program counts between variations #2, #3, and #4; Test type: Superiority; p = 0.017, Chi-squared; Total Count - Cramer's V = 0.45
Statistical Analysis 5: Comparison: Participants With Hearing Loss; This is to see if there is a difference in somewhat preferred (i.e. rated in the middle) program counts between variations #2 and #3; Test type: Superiority; p = 0.02, Chi-squared; Total Count - Cramer's V = 0.51
Statistical Analysis 6: Comparison: Participants With Hearing Loss; This is to see if there is a difference in somewhat preferred (i.e. rated in the middle) program counts between variations #2 and #4; Test type: Superiority; p = 0.006, Chi-squared; Total Count - Cramer's V = 0.61
Statistical Analysis 7: Comparison: Participants With Hearing Loss; This is to see if there is a difference in the least preferred program counts between variations #2, #3, and #4; Test type: Superiority; p < .0001, Chi-squared; Total Count - Cramer's V = 0.6
Statistical Analysis 8: Comparison: Participants With Hearing Loss; This is to see if there is a difference in the least preferred program counts between variations #2 and #3; Test type: Superiority; p = 0.08, Chi-squared; Total Count - Cramer's V = 0.38
Statistical Analysis 9: Comparison: Participants With Hearing Loss; This is to see if there is a difference in the least preferred program counts between variations #2 and #4; Test type: Superiority; p < 0.001, Chi-squared; Total Count - Cramer's V = 0.5

ADVERSE EVENTS:
Time Frame: Participants were exposed to multiple interventions at once and had the ability to cycle through the various interventions (frequency curves). For this reason, adverse event data would have been collected per task and not intervention due to the quick exposure to multiple interventions. Adverse Event Data per participant was collected and is reported below. Sound Quality Ratings - Live - 2 hours Sound Quality Ratings - Streaming - 1 hour US Matrix Test Task - 30 minutes
Groups:
- Participants With Hearing Loss - Sound Quality Ratings Task - Live; Participants With Hearing Loss - Sound Quality Ratings Task - Streaming; Participants With Hearing Loss - US Matrix Test Task: Individuals with hearing loss that meet the candidacy to wear hearing aids. All interventions are associated with the fitting of binaural hearing aids with various coupling methods. All participants will be assessed under all interventions.
  Interventions each participant was exposed to:
  Standard Curve under Program 1
  Variation #1 under Program 1
  Standard Curve under Program 2
  Variation #1 under Program 2
  Standard Curve under Program 3
  Variation #1 under Program 3
  Standard Curve under Program 4
  Variation #1 under Program 4
  Variation #2 under Program 5 - Streaming Only
  Variation #3 under Program 5 - Streaming Only
  Variation #4under Program 5 - Streaming Only
  Unaided
Arm/Group | Participants With Hearing Loss - Sound Quality Ratings Task - Live | Participants With Hearing Loss - Sound Quality Ratings Task - Streaming | Participants With Hearing Loss - US Matrix Test Task
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-07-24): https://cdn.clinicaltrials.gov/large-docs/17/NCT05828017/Prot_SAP_000.pdf